CLINICAL TRIAL: NCT00731029
Title: Comparative Vaccination Study of the Reactogenicity and Immunogenicity of a Thiomersal-Free Formulation of Influsplit SSW® 2002/2003 Versus the Standard Formulation of Influsplit SSW® 2002/2003 in Individuals Over 18 Years
Brief Title: Reacto & Immunogenicity of TF Formulation of Influsplit SSW® 2002/03 v/s Std Formulation of Influsplit SSW® 2002/03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK Biologicals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 218352/053
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Influenza
Keywords: Influenza; Thiomersal-free influenza split vaccine 2002/2003; Influsplit SSW®/Fluarix™ 2002/2003
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group A (Experimental): The subjects in this group will be 18-60 years.
  Interventions: Biological: Thiomersal free trivalent influenza split vaccine 2002/2003
- Group B (Experimental): The subjects in this group will be > 60 years.
  Interventions: Biological: Thiomersal free trivalent influenza split vaccine 2002/2003
- Group C (Active Comparator): The subjects in this group will be 18-60 years.
  Interventions: Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2002/2003
- Group D (Active Comparator): The subjects in this group will be > 60 years.
  Interventions: Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2002/2003

INTERVENTIONS:
Biological: Thiomersal free trivalent influenza split vaccine 2002/2003 — Single dose, intramuscular injection
  Arms: Group A; Group B
Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2002/2003 — Single dose, intramuscular injection
  Arms: Group C; Group D

SUMMARY:
This is a comparative vaccination study of the reactogenicity and immunogenicity of a thiomersal-free formulation of Influsplit SSW® 2002/2003 versus the standard formulation of Influsplit SSW® 2002/2003 in individuals over 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who are capable of being vaccinated and subjects with primary diseases (cardiovascular conditions, metabolic conditions such as diabetes mellitus, respiratory diseases) who are capable of being vaccinated and aged over 18 years who want to be vaccinated against influenza or for whom the doctor considers prophylactic influenza immunisation to be indicated.
* The inclusion of individuals who had not been immunised in the 2001/2002 season is preferred.
* Written consent to vaccination must be available after the subjects have been briefed on the study in understandable language.

Exclusion Criteria:

* Use of study or unlicensed medication or administration of a vaccine other than the study vaccine within 30 days preceding vaccination and/or during the study period
* Acute disease at the beginning of the study
* Acute clinically significant changes in the lungs, cardiovascular system, liver or kidney function, identified by physical examination or laboratory tests
* Pregnancy
* Women who would like to fall pregnant during the period from the day of vaccination to 1 month thereafter
* Known allergic reactions that might have been caused by one or more ingredients of the vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2002-09; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
GMT of the haemagglutination-inhibiting antibodies (HIA) and calculation of seroconversion factor, seroconversion rate and seroprotection rate checked against the CHMP criteria. The seroprotection power will be calculated as well. | On Day 21 (± 2) after vaccination
Descriptive comparison of the occurrence, severity and causal relationship to vaccination of solicited local and general symptoms | Within 4 days after vaccination

SECONDARY OUTCOMES:
Descriptive comparison of the occurrence and causal relationship to vaccination of unsolicited signs and symptoms | Within 30 days after vaccination
Descriptive comparison of the occurrence, severity and causal relationship to vaccination of any serious adverse events (SAEs) | During the entire study period.
Investigation of antibody persistence assessed by the criteria of the CHMP. | 11, 19, 27 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Dresden, Germany